CLINICAL TRIAL: NCT02223637
Title: MENVEO Pregnancy Registry: an Observational Study on the Safety of MENVEO Exposure in Pregnant Women and Their Offspring
Brief Title: Meningococcal Quadrivalent CRM-197 Conjugate Vaccine Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 205531; V59_72OB (Other: Novartis)
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-03

CONDITIONS: Meningococcal Disease; Pregnancy; Infections, Meningococcal
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months

GROUPS / COHORTS (1):
- Exposure group: Pregnant women who were exposed to
  ≥1 dose of Menveo vaccine within 28 days prior to conception or at any time during pregnancy were included.
  Interventions: Biological: Meningococcal quadrivalent CRM-197 conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal quadrivalent CRM-197 conjugate vaccine — This pregnancy registry is strictly observational. Decisions of vaccination are made by health care providers.

SUMMARY:
The GlaxoSmithKline's Meningococcal quadrivalent CRM-197 conjugate vaccine pregnancy registry is established to meet a post marketing commitment agreed upon with CBER to prospectively collect data on pregnancy exposures to Meningococcal quadrivalent CRM-197 conjugate vaccine.

It is an observational study of women inadvertently immunized with the Meningococcal quadrivalent CRM-197 conjugate vaccine within 28 days prior to conception or at any time during pregnancy as part of routine care.

The objective of the pregnancy registry is to evaluate pregnancy outcomes among women immunized with the Meningococcal quadrivalent CRM-197 conjugate vaccine within 28 days prior to conception or at any time during pregnancy. The primary outcomes of interest include major congenital malformation, preterm birth, and low birth weight. Other pregnancy outcomes will be collected, including spontaneous abortions and stillbirths.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient evidence to confirm that MENVEO exposure occurred within 28 days prior to conception or at any time during pregnancy
* Sufficient information to determine whether the pregnancy is prospectively or retrospectively registered (ie, whether the outcome of pregnancy was known at the time of first contact with the registry)
* Date the pregnancy exposure is registered
* Full reporter (ie, HCP) contact information to allow for follow-up (name, address, etc.)

Exclusion Criteria:

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include pregnant women within the United States who were immunized with the GlaxoSmithKline's Meningococcal quadrivalent CRM-197 conjugate vaccine within 28 days prior to conception or at any time during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilmington, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 93 subjects included in the registry,82 subjects were included for analysis as 7 lost to follow up & 4 were invalid cases. Of these 82 subjects,1 pregnancy resulted in 1 set of twins birth.Analyses on outcome measures were performed on pregnant outcomes(Analysis population pregnancy outcomes)& on live births(Analysis population live births)
Period: Overall Study
Arm/Group | Exposure Group
Started | 82
Completed | 82
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exposure Group
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: Months] | 18.9 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race - White or Caucasian | 14
  Race - Black or African American | 12
  Race - Asian | 1
  Race - Native Hawaiian or Other Pacific Islander | 2
  Race - Other | 52
  Race - Unknown | 1
  Ethnicity - Hispanic or Latino | 57
  Ethnicity - Not Hispanic or Latino | 23
  Ethnicity - Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Live Births Reported With Major Congenital Malformations (MCM) on Exposure to Menveo Within 28 Days Prior to Conception
Description: The pregnancy registry defined an MCM as any major structural or chromosomal defect or combination of 2 or more conditional defects in live-born infants, stillbirths, or fetal losses of any gestational age. This outcome measure was analyzed on live births reported with MCM, for subjects who were exposed to Menveo vaccine within 28 days prior to conception. The prevalence estimate of MCM was calculated as proportions of live births with MCM from the total number of live births
Time Frame: From the time of enrolment until the date of pregnancy outcome documentation (i.e. From registration upon Menveo exposure within 28 days prior to conception until the estimated delivery date)
Population: The analysis was performed on live births who were exposed to Menveo vaccine within 28 days prior to conception
Measure: Number; unit: Percentage of Live Births with MCM
Groups:
- Live Births Group: All live births (single or multiple) who were exposed to Menveo vaccine within 28 days prior to conception or at any time during the mother's pregnancy
Arm/Group | Live Births Group
Number analyzed (Participants) | 13
Percentage of Live Births with MCM
  Live births with MCM | 0.0
  Live births without MCM | 84.6
  Live births with no known defects | 15.4

2. Primary Outcome: Percentage of Live Births Reported With Major Congenital Malformations (MCM) on Exposure to Menveo Vaccine During the First Trimester
Description: The pregnancy registry defined an MCM as any major structural or chromosomal defect or combination of 2 or more conditional defects in live-born infants, stillbirths, or fetal losses of any gestational age. This outcome measure was analyzed on live births reported with MCM, for subjects who were exposed to Menveo vaccine during the first trimester of pregnancy.The prevalence estimate of MCM was calculated as proportions of live births with MCM from the total number of live births.
Time Frame: From the time of enrolment until the date of pregnancy outcome documentation (i.e.From registration upon Menveo exposure during first trimester of pregnancy [0-13 weeks] until the estimated delivery date)
Population: The analysis was performed on live births who were exposed to Menveo vaccine during the first trimester of pregnancy
Measure: Number; unit: Percentage of Live Births with MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 39
Percentage of Live Births with MCM
  Live births with MCM | 2.6
  Live births without MCM | 87.2
  Live births with no known defects | 10.3

3. Primary Outcome: Percentage of Live Births Reported With Major Congenital Malformations (MCM) on Exposure to Menveo Vaccine During the Second Trimester
Description: The pregnancy registry defined an MCM as any major structural or chromosomal defect or combination of 2 or more conditional defects in live-born infants, stillbirths, or fetal losses of any gestational age. This outcome measure was analyzed on live births reported with MCM, for subjects who were exposed to Menveo vaccine during the second trimester of pregnancy.The prevalence estimate of MCM was calculated as proportions of live births with MCM from the total number of live births
Time Frame: From the time of enrolment until the date of pregnancy outcome documentation (i.e. from registration upon Menveo exposure during second trimester of pregnancy [14-27 weeks] until the estimated delivery date)
Population: The analysis was performed on live births who were exposed to Menveo vaccine during second trimester of pregnancy
Measure: Number; unit: Percentage of Live Births with MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 2
Percentage of Live Births with MCM
  Live births with MCM | 50.0
  Live births without MCM | 50.0
  Live births with no known defects | 0.0

4. Primary Outcome: Percentage of Live Births Reported With Major Congenital Malformations (MCM) on Exposure to Menveo Vaccine During Third Trimester
Description: The pregnancy registry defined an MCM as any major structural or chromosomal defect or combination of 2 or more conditional defects in live-born infants, stillbirths, or fetal losses of any gestational age. This outcome measure was analyzed on live births reported with MCM, for subjects who were exposed to Menveo vaccine during the third trimester of pregnancy.The prevalence estimate of MCM was calculated as proportions of live births with MCM from the total number of live births
Time Frame: From the time of enrolment until the date of pregnancy outcome documentation (i.e.From registration upon Menveo exposure during third trimester of pregnancy [>27 weeks] until the estimated delivery date)
Population: The analysis was performed on live births who were exposed to Menveo vaccine during third trimester of pregnancy
Measure: Number; unit: Percentage of Live Births with MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 1
Percentage of Live Births with MCM
  Live births with MCM | 0.0
  Live births without MCM | 100.0
  Live births with no known defects | 0.0

5. Primary Outcome: Percentage of Live Births Reported With Major Congenital Malformations (MCM) on Exposure to Menveo Within 28 Days Prior to Conception or at Any Time During the Pregnancy
Description: The pregnancy registry defined an MCM as any major structural or chromosomal defect or combination of 2 or more conditional defects in live-born infants, stillbirths, or fetal losses of any gestational age. This outcome measure was analyzed on live births reported with MCM, for subjects who were exposed to Menveo vaccine within 28 days prior to conception or at any time during the pregnancy.The prevalence estimate of MCM was calculated as proportions of live births with MCM from the total number of live births
Time Frame: From the time of enrolment until the date of pregnancy outcome documentation (i.e. from registration upon exposure to Menveo within 28 days prior to conception or at any time during pregnancy until the estimated delivery date)
Population: The analysis was performed on live births who were exposed to Menveo vaccine within 28 days prior to conception or at any time during the pregnancy
Measure: Number; unit: Percentage of Live Births with MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 55
Percentage of Live Births with MCM
  Live births with MCM | 3.6
  Live births without MCM | 85.5
  Live births with no known defects | 10.9

6. Primary Outcome: Percentage of Preterm Births Reported on Exposure to Menveo Vaccine Within 28 Days Prior to Conception
Description: A pregnancy outcome that is reported with a preterm birth represents an infant born at a gestational age under (<) 37 weeks. The prevalence rate of preterm birth was calculated as a proportion, with the number of preterm births as the numerator and the number of live births as the denominator. Because MCMs are often associated with preterm birth and LBW, infants with MCMs were excluded from analyses of this outcome measure and were not counted in the numerator or denominator when prevalence rate was determined.
Time Frame: as for outcome 1
Population: The analysis was performed on live births who were exposed to Menveo vaccine within 28 days prior to conception
Measure: Number; unit: Percentage of preterm births without MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 13
Percentage of preterm births without MCM | 23.1

7. Primary Outcome: Percentage of Preterm Births Reported on Exposure to Menveo Vaccine During the First Trimester
Description: as for outcome 6
Time Frame: From the time of enrolment until the date of pregnancy outcome documentation (i.e. from registration upon Menveo exposure during first trimester of pregnancy [0-13 weeks] until the estimated delivery date)
Population: The analysis was performed on the live births who were exposed to Menveo vaccine during the first trimester of pregnancy
Measure: Number; unit: Percentage of preterm births without MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 38
Percentage of preterm births without MCM | 10.5

8. Primary Outcome: Percentage of Preterm Births Reported on Exposure to Menveo Vaccine During the Second Trimester
Description: as for outcome 6
Time Frame: as for outcome 3
Population: The analysis was performed on the live births who were exposed to Menveo vaccine during the second trimester of pregnancy
Measure: Number; unit: Percentage of preterm births without MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 1
Percentage of preterm births without MCM | 100.0

9. Primary Outcome: Percentage of Preterm Births Reported on Exposure to Menveo Vaccine During the Third Trimester
Description: as for outcome 6
Time Frame: From the time of enrolment until the date of pregnancy outcome documentation (i.e. from registration upon Menveo exposure during third trimester of pregnancy (>27 weeks) until the estimated delivery date)
Population: The analysis was performed on the live births who were exposed to Menveo vaccine during the third trimester of pregnancy
Measure: Number; unit: Percentage of preterm births without MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 1
Percentage of preterm births without MCM | 0.0

10. Primary Outcome: Percentage of Preterm Births Reported on Exposure to Menveo Vaccine Within 28 Days Prior to Conception or at Any Time During the Pregnancy
Description: as for outcome 6
Time Frame: as for outcome 5
Population: The analysis was performed on the live births who were exposed to Menveo vaccine within 28 days prior to conception or at any time during the mother's pregnancy
Measure: Number; unit: Percentage of preterm births without MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 53
Percentage of preterm births without MCM | 15.1

11. Primary Outcome: Percentage of Low Birth Weight (LBW) Live Births Reported on Exposure to Menveo Vaccine Vaccine Within 28 Days Prior to Conception
Description: A pregnancy outcome that is reported as a LBW birth represents an infant whose birth weight is <2500 g. The prevalence rate of LBW was calculated as a proportion, with the number of LBW infants as the numerator and the number of live births as the denominator. Infants with MCMs were excluded from the analysis of this outcome measure as MCMs are often associated with LBW.
Time Frame: as for outcome 1
Population: The analysis was performed on live births who were exposed to Menveo vaccine within 28 days prior to conception
Measure: Number; unit: Percentage of LBW live birth without MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 13
Percentage of LBW live birth without MCM | 15.4

12. Primary Outcome: Percentage of LBW Live Births Reported on Exposure to Menveo Vaccine During the First Trimester
Description: as for outcome 11
Time Frame: as for outcome 7
Population: The analysis was performed on live births who were exposed to Menveo vaccine during the first trimester of pregnancy
Measure: Number; unit: Percentage of LBW live birth without MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 38
Percentage of LBW live birth without MCM | 5.3

13. Primary Outcome: Percentage of LBW Live Births Reported on Exposure to Menveo Vaccine During the Second Trimester
Description: as for outcome 11
Time Frame: as for outcome 3
Population: as for outcome 8
Measure: Number; unit: Percentage of LBW live birth without MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 1
Percentage of LBW live birth without MCM | 100.0

14. Primary Outcome: Percentage of LBW Live Births Reported on Exposure to Menveo Vaccine During the Third Trimester
Description: as for outcome 11
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number; unit: Percentage of LBW live birth without MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 1
Percentage of LBW live birth without MCM | 0.0

15. Secondary Outcome: Number of Pregnancy Outcomes Reported for Subjects Exposed to Menveo Within 28 Days Prior to Conception
Description: The pregnancy outcomes assessed were: live births, stillbirths, SABs, IABs, ectopic pregnancy, molar pregnancy and others.
  Spontaneous abortions (SABs) are defined as fetal death or expulsion of products of conception prior to 20 weeks gestation.
  Induced abortions (IABs) are defined as voluntary interruption of pregnancy, including pregnancy termination that occurs electively, to preserve maternal health, or due to fetal abnormalities.
  Stillbirths are defined as fetal death occurring at 20 weeks gestation or greater, or if gestation age is unknown, a fetus weighing 500 g or more.
  Ectopic pregnancy is defined as implantation of a conception outside of the uterus.
  Molar pregnancy is defined as a conception that results in a gestational trophoblastic tumor.
Time Frame: as for outcome 1
Population: The analysis was performed on subjects who were exposed to Menveo vaccine within 28 days prior to conception
Measure: Number; unit: Pregnancy outcomes
Arm/Group | Exposure Group
Number analyzed (Participants) | 16
Pregnancy outcomes
  Live Births | 12
  Stillbirth | 0
  SAB | 2
  IAB | 2
  Ectopic pregnancy | 0
  Molar pregnancy | 0
  Others | 0

16. Secondary Outcome: Number of Pregnancy Outcomes Reported for Subjects Exposed to Menveo During the First Trimester
Description: The pregnancy outcomes assessed were: live births, stillbirths, SABs, IABs, ectopic pregnancy, molar pregnancy and others.
Time Frame: as for outcome 7
Population: The analysis was performed on subjects who were exposed to Menveo vaccine during the first trimester of pregnancy
Measure: Number; unit: Pregnancy outcomes
Arm/Group | Exposure Group
Number analyzed (Participants) | 59
Pregnancy outcomes
  Live Births | 39
  Stillbirths | 0
  SAB | 7
  IAB | 13
  Ectopic pregnancy | 0
  Molar pregnancy | 0
  Others | 0

17. Secondary Outcome: Number of Pregnancy Outcomes Reported for Subjects Exposed to Menveo Vaccine During the Second Trimester
Description: The pregnancy outcomes assessed were: live births, stillbirths, SAB, IAB, ectopic pregnancy, molar pregnancy and others
Time Frame: as for outcome 3
Population: The analysis was performed on subjects who were exposed to Menveo vaccine during the second trimester of pregnancy
Measure: Number; unit: Pregnancy outcomes
Arm/Group | Exposure Group
Number analyzed (Participants) | 2
Pregnancy outcomes
  Live Births | 2
  Stillbirths | 0
  SAB | 0
  IAB | 0
  Ectopic pregnancy | 0
  Molar pregnancy | 0
  Others | 0

18. Secondary Outcome: Number of Pregnancy Outcomes Reported for Subjects Exposed to Menveo Vaccine During the Third Trimester
Description: The pregnancy outcomes assessed were: Live births, stillbirths, SAB,IAB, ectopic pregnancy, molar pregnancy and others.
Time Frame: as for outcome 9
Population: The analysis was performed on subjects who were exposed to Menveo vaccine during the third trimester of pregnancy
Measure: Number; unit: Pregnancy outcomes
Arm/Group | Exposure Group
Number analyzed (Participants) | 1
Pregnancy outcomes
  Live Births | 1
  Stillbirths | 0
  SAB | 0
  IAB | 0
  Ectopic pregnancy | 0
  Molar pregnancy | 0
  Others | 0

19. Secondary Outcome: Number of Pregnancy Outcomes Reported for Subjects Exposed to Menveo Vaccine Within 28 Days Prior to Conception or at Any Time During the Pregnancy
Description: The pregnancy outcomes assessed were: Live births,stillbirths, SAB, IAB, ectopic pregnancy, molar pregnancy and others.
Time Frame: as for outcome 5
Population: The analysis was performed on subjects who were exposed to Menveo vaccine within 28 days prior to pregnancy or at any time during the pregnancy.
Measure: Number; unit: Pregnancy outcomes
Arm/Group | Exposure Group
Number analyzed (Participants) | 82
Pregnancy outcomes
  Live Births | 54
  Stillbirths | 0
  SAB | 10
  IAB | 18
  Ectopic pregnancy | 0
  Molar pregnancy | 0
  Others | 0

20. Primary Outcome: Percentage of LBW Live Births Reported on Exposure to Menveo Vaccine Within 28 Days Prior to Conception or at Any Time During the Pregnancy
Description: as for outcome 11
Time Frame: as for outcome 5
Population: The analysis was performed on the live births who were exposed to Menveo vaccine within 28 days prior to conception or at any time during the pregnancy
Measure: Number; unit: Percentage of LBW live birth without MCM
Arm/Group | Live Births Group
Number analyzed (Participants) | 53
Percentage of LBW live birth without MCM | 9.4

ADVERSE EVENTS:
Time Frame: No adverse events data was collected in this study.
Description: No adverse events data was collected in this study.
Arm/Group | Exposure Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trials.

DOCUMENTS (2):
  • Study Protocol (2014-09-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT02223637/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT02223637/SAP_001.pdf